CLINICAL TRIAL: NCT04896112
Title: An Open-Label, Multicenter, Phase I Study to Evaluate the Safety, Pharmacokinetics and Preliminary Efficacy of LNK01002 in Patients With Malignant Myeloid Hematologic Neoplasms
Brief Title: A Study of LNK01002 in Patients With Primary or Secondary Myelofibrosis,Polycythemia Vera or Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Lynk Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LNK-1002-01; IND 153144 (Registry Identifier: FDA)
Record Dates: First submitted 2021-05-08; First posted 2021-05-21 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Acute Myeloid Leukemia; Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Polycythemia Vera
Keywords: Malignant Myeloid Hematologic Neoplasms; Primary Myelofibrosis; Post-polycythemia Vera Myelofibrosis; Post-essential Thrombocythemia Myelofibrosis; Myeloid malignancies; Myelofibrosis; Polycythemia Vera; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Primary Myelofibrosis; Polycythemia Vera

STUDY DESIGN:
Intervention Model Description: An Open-Label, Multicenter, Phase I Study to Evaluate the Safety, Pharmacokinetics and Preliminary Efficacy of LNK01002
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Patient with Malignant Myeloid Hematologic Neoplasms treated with LNK01002 15 mg (Experimental): Single dose of LNK01002 15 mg; followed by a 3-day observation period then 15mg BID in 28-day treatment cycles
  Interventions: Drug: LNK01002
- Patients with Malignant Myeloid Hematologic Neoplasms treated with LNK01002 30 mg (Experimental): LNK01002 30 mg twice daily (BID), followed by a 3-day observation period then 30 mg BID in 28-day treatment cycles
  Interventions: Drug: LNK01002
- Patients with Malignant Myeloid Hematologic Neoplasms treated with LNK01002 60 mg (Experimental): LNK01002 60 mg BID, followed by a 3-day observation period then 60 mg BID in 28-day treatment cycles
  Interventions: Drug: LNK01002
- Patients with Malignant Myeloid Hematologic Neoplasms treated with LNK01002 100 mg (Experimental): LNK01002 100 mg BID, followed by a 3-day observation period then 100 mg BID in 28-day treatment cycles
  Interventions: Drug: LNK01002
- Patients with Malignant Myeloid Hematologic Neoplasms treated with LNK01002 150 mg (Experimental): LNK01002 150 mg BID, followed by a 3-day observation period then 150 mg BID in 28-day treatment cycles
  Interventions: Drug: LNK01002
- Patients with Malignant Myeloid Hematologic Neoplasms treated with LNK01002 200 mg (Experimental): LNK01002 200 mg BID, followed by a 3-day observation period then 200 mg BID in 28-day treatment cycles
  Interventions: Drug: LNK01002
- Patients with Malignant Myeloid Hematologic Neoplasms treated with LNK01002 260 mg (Experimental): LNK01002 260 mg BID, followed by a 3-day observation period then 260 mg BID in 28-day treatment cycles
  Interventions: Drug: LNK01002
- Patients with Acute Myeloid Leukemia With Mutant FLT3 (Experimental): LNK01002 at the RP2D dose in 28-day treatment cycles
  Interventions: Drug: LNK01002
- Patients with Malignant Myeloid Hematologic Neoplasms Without Mutant FLT3 (Experimental): LNK01002 at the RP2D dose in 28-day treatment cycles
  Interventions: Drug: LNK01002
- Patients with Primary or Secondary Myelofibrosis,PV (Experimental): LNK01002 at the RP2D dose in 28-day treatment cycles
  Interventions: Drug: LNK01002

INTERVENTIONS:
Drug: LNK01002 — LNK01002 will be administrated orally.
  Other Names: LNK-1000318

SUMMARY:
This multicenter, open-label, phase 1 study designed to evaluate safety and tolerability of multi-kinase inhibitor LNK01002 in patients with primary myelofibrosis (PMF), or MF due to polycythemia vera (PV-MF), or essential thrombocythemia (ET-MF), polycythemia vera (PV), or with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-finding study of the triple kinase inhibitor LNK01002 in patients with Malignant Myeloid Hematologic Neoplasms. The study consists of two periods: the dose escalation, main period and a dose expansion period. In the dose escalation period, successive cohorts of patients with Malignant Myeloid Hematologic Neoplasms will be enrolled to establish the maximum tolerated dose. In the dose expansion period (dose-confirmation phase), three cohorts of patients will be enrolled: AML patients with confirmed FLT3-ITD mutations, AML patients without FLT3-ITD mutations, and patients with primary MF ,PV or PV/ET-MF.

The safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary clinical activity of LNK01002 in patients with Malignant Myeloid Hematologic Neoplasms will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years old or older, male or female.
2. Patients must have histologically or cytologically confirmed tumors of the following types.

   * Dose Escalation Phase: Patients with PMF,PV/ET-MF,PV

     1. Intermediate or high-risk primary myelofibrosis, intermediate or high-risk post-polycythemia vera myelofibrosis , or post-essential thrombocythemia myelofibrosis , or high-risk polycythemia vera who have no available therapy or relapsed after allogeneic hematopoietic cell transplantation.
     2. Symptomatic splenomegaly
     3. Not undergone splenectomy or splenic radiation therapy within 6 months prior to screening.
   * Dose expansion phase: Patients with PMF, PV/ET-MF,PV who relapsed or are intolerant to standard treatment, and relapsed/refractory AML
3. Platelet count ≥ 100 × 10e9/L within 14 days before study drug administration
4. Absolute neutrophil count (ANC) ≥ 1.5 × 10e9/L within 14 days before study drug administration
5. Women of childbearing potential negative pregnancy test at screening. Female patients of childbearing potential, or male patients and their partners should agree to effective contraception from signing ICF until 6 months after the last dose of study drug.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria will be excluded from the clinical study:

1. Allergic to any component of LNK01002.
2. Serum total bilirubin greater than 1.5 times the upper limit of the normal (ULN) reference range, except patients diagnosed as Gilbert's disease
3. ALT or AST higher than 3 times the ULN reference range without hepatic involvement by leukemia, which are excluded if higher than 5 times the ULN
4. Glomerular filtration rate or estimated creatinine clearance < 50 mL/min according to the Cockcroft-Gault formula;
5. Serum amylase or lipase levels higher than the ULN and considered clinically significant
6. International normalized ratio (INR) or partial activated prothrombin time (aPTT) above 1.5 times the ULN reference range
7. Known history of clinically significant liver disease, including viral or other hepatitis:

   a) Patients with hepatitis B or hepatitis C may be enrolled if they have a negative polymerase chain reaction (PCR)
8. Known human immunodeficiency virus (HIV) infection;
9. Clinically significant cardiovascular diseases, including acute myocardial infarction, unstable angina, coronary artery bypass surgery within 6 months before enrollment, congestive heart failure with New York Heart Association (NYHA) classification of III or above, left ventricular ejection fraction (LVEF) < 50%, or uncontrolled hypertension, cardiac arrhythmia;
10. Patients with history or presence of clinically relevant non-malignant CNS disease requiring treatment;
11. Patients who have received systemic antineoplastic therapy or radiotherapy within 2 weeks prior to start of study treatment;
12. Patients who have received hematopoietic stem cell transplantation (HSCT) within 60 days prior to the start of study treatment, or are receiving immunosuppressive therapy after HSCT at screening, or have graft-versus-host disease (GVHD) requiring ongoing treatment;
13. Received anti-tumor Chinese herbal medicine treatment within 1 week before the start of study treatment;
14. Received CYP3A strong inhibitors or strong inducers less than one week or 5 half-lives (whichever is longer) prior to the start of study treatment;
15. Uncontrolled, active infections requiring intravenous antibiotic treatment;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Assessing the safety and tolerability of LNK01002 in patients with Malignant Myeloid Hematologic Neoplasms | 31 days
  Assessed by monitoring the frequency, duration and severity of adverse events and serious adverse events.
Assessing maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of LNK01002 in patients with Malignant Myeloid Hematologic Neoplasms | 31 days
  Maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) will be assessed based on the safety profile by the SRC
Assessing the preliminary antitumor activity of LNK01002 | 24 Weeks
  The preliminary antitumor activity will be analyzed in patients with different types of malignant myeloid hematologic neoplasms by response rate using bone marrow and hematologic analyses (MF/AML) or by the MF Symptom Assessment Scale and spleen volume by MRI (MF).

SECONDARY OUTCOMES:
Measurement of pharmacokinetic (PK) parameter, AUC, in MF, PV,PV-MF or ET-MF patients | Day 1, Day 2, and Day 15
  Measurement will be using extensive PK sampling
Measurement of pharmacokinetic (PK) parameter, Cmax, in MF, PV,PV-MF or ET-MF patients | Day 1, Day 2, and Day 15
  Measurement will be using extensive PK sampling
Measurement of pharmacokinetic (PK) parameter, Tmax, in MF, PV, PV-MF or ET-MF patients | Day 1, Day 2, and Day 15
  Measurement will be using extensive PK sampling
Measurement of pharmacokinetic (PK) parameter, CL/F, in MF, PV, PV-MF or ET-MF patients | Day 1, Day 2, and Day 15
  Measurement will be using extensive PK sampling
Measurement of pharmacokinetic (PK) parameter, T1/2, in MF, PV, PV-MF or ET-MF patients | Day 1, Day 2, and Day 15
  Measurement will be using extensive PK sampling
Measurement of pharmacokinetic (PK) parameter, Vz/F, in MF, PV,PV-MF or ET-MF patients | Day 1, Day 2, and Day 15
  Measurement will be using extensive PK sampling
Measurement of pharmacokinetic (PK) parameter, MRT, in MF, PV,PV-MF or ET-MF patients | Day 1, Day 2, and Day 15
  Measurement will be using extensive PK sampling

CONTACTS AND LOCATIONS:
Overall Officials: Linda Wei, M.D., Study Director — Lynk Pharmaceuticals Co., Ltd
Locations (2):
- United States (2):
  - Revive Research Institute, Farmington Hills, Michigan
  - Revive Research Institute, Sterling Heights, Michigan

IPD SHARING:
Plan to Share IPD: No